CLINICAL TRIAL: NCT06090630
Title: Non-Uniformly Sampled MR Correlated Spectroscopic Imaging in Breast Cancer and Nonlinear Reconstruction
Brief Title: MR Correlated Spectroscopic Imaging for Diagnosing Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-000933; NCI-2019-02258 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-07

CONDITIONS: Benign Breast Neoplasm; Breast Carcinoma; Malignant Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (DWI, magnetic resonance spectroscopic imaging) (Experimental): Participants undergo DWI over 15 minutes and MR spectroscopic imaging over 45 minutes.
  Interventions: Procedure: Diffusion Weighted Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging

INTERVENTIONS:
Procedure: Diffusion Weighted Imaging — Undergo DWI-MRI
  Other Names: Diffusion Weighted MRI; Diffusion-Weighted Magnetic Resonance Imaging; Diffusion-Weighted MR Imaging; Diffusion-Weighted MRI; DW-MRI; DWI; DWI MRI; DWI-MRI; MR Diffusion-Weighted Imaging
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MR spectroscopic imaging
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; MS; Proton Magnetic Resonance Spectroscopic Imaging

SUMMARY:
This trial studies how well an imaging technique called magnetic resonance (MR) spectroscopic imaging works in identifying breast cancer in women with benign or suspicious areas in the breast. Magnetic resonance imaging (MRI) is a diagnostic tool used to investigate the location of tumors in different organs. Since radiological pictures do not have sufficient information for tumor grades, invasive procedure such as biopsy is performed on patients with breast cancers for diagnosis. Breast tissue contains water, fat, and chemicals known as metabolites. MR spectroscopic imaging may help to characterize the various breast metabolite steady state levels and identify the differences between necrosis and tumor recurrence, which is difficult using radiological procedures such as MRI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Non-uniform undersampling schemes (NUS) will be combined with 5-dimensional (5D) echo-planar imaging based correlated spectroscopic imaging (EP-COSI) sequence.

II. Group sparsity (GS)-based compressed-sensing (CS) reconstruction schemes will be developed for accelerated acquisition and optimized to reconstruct the NUS EP-COSI data with better reliability.

III. Alterations in metabolite and lipid levels will be correlated with apparent diffusion coefficient (ADC) changes in breast cancer patients compared to healthy women which will improve the diagnostic accuracy.

OUTLINE:

Participants undergo diffusion weighted imaging (DWI)-MRI over 15 minutes and MR spectroscopic imaging over 45 minutes.

After completion of study, participants are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Malignant tumor subjects must have malignant needle biopsy results with concordant imaging and pathological findings.
* Benign tumor subjects must have benign needle biopsy results. Benign subjects will only include those with concordant benign imaging and pathological findings.
* Control subjects: healthy and have no previous history of any type of cancers.
* The women should be able to read and understand English. Hence, non-English speaking subjects will be excluded. However, if there will be a necessity of translating the written informed consent form in the subject's mother tongue (such as Hispanic, Chinese, Persian, Indian, etc.), the translated consent form will be submitted for expedited approval to the office of University of California, Los Angeles (UCLA) Institutional Review Board (IRB).

Exclusion Criteria:

* Pregnant women will be excluded.
* Breast feeding women.
* MR incompatible items: cardiac pacemaker, aneurysm clip, heart valve prosthesis, nitroglycerin transdermal patch, implanted cardiac defibrillator, implanted electrode, including pacing wires, cochlear implant, other, implanted drug infusion device, implanted insulin pump, intravascular coil, filter or stent: (e.g., Gianturco coil, Gunther inferior vena cava [IVC] filter, etc.), intraventricular shunt, neurostimulator/biostimulator, Swan-Ganz catheter, any type of electronic, mechanical or magnetic implant, any type of implant held in place by a magnet, artificial limb or joint, contraceptive device (e.g., intrauterine device [IUD], diaphragm), dentures, ear implant, eye/orbital implant, foreign body (e.g., shrapnel, bullet, etc.), halo vest or metallic cervical fixation device, orthopedic item (for example: pins, rods, screws, clips, plates, wires, etc.), surgical clip or staple, vascular access port, wire mesh, hearing aid (must remove prior to the exam), tattooed eyeliner (a small percentage of patients with tattooed eyeliner have experienced transient skin irritation in association with MRI). The patients using transdermal patches will be asked to remove the patch and will be excluded if the patch cannot be removed.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Apparent diffusion coefficient (ADC) maps | At the time of imaging
  ADC maps will be calculated from diffusion weighted (DW) images by using linear regression of logarithmic intensities by using software for combinations of two, three, four, and five DW images with different b values. ADC maps will also be calculated for the remaining combinations of up to 10 evenly distributed b values. In total, 501 value combinations will be automatically processed and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Thomas, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States